CLINICAL TRIAL: NCT04738136
Title: A Randomized, Open-Label, Controlled, Phase II Study to Evaluate the Safety, Tolerability and Efficacy Of S-1226 In Hospitalized Subjects With Moderate Severity Covid-19 Bronchiolitis/Pneumonia
Brief Title: Safety, Tolerability and Efficacy Of S-1226 in Moderate Severity Covid-19 Bronchiolitis/Pneumonia
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: SolAeroMed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAMi-05-1-01
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-02

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: S-1226; Moderate Severity Covid-19 infection; SolAeroMed; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — perfluorooctylbromide and CO2 drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Subjects will only receive standard of care treatment for moderate severity COVID19 bronchiolitis/pneumonia.
- Standard of Care(SOC) + S-1226 at either 4% 8% or 12% CO2 (Experimental): Subjects will receive SOC plus the highest tolerated dose of S-1226 at either 4% 8% or 12% CO2 twice daily for up to 5 consecutive days.
  Interventions: Drug: S-1226

INTERVENTIONS:
Drug: S-1226 — S-1226 has two components delivered by inhalation. It is a mixture of perfluorooctylbromide (PFOB) delivered in vapour form within a medical gas mixture containing CO2. The PFOB component remains the same but the medical gas component contains 4%, 8%, or 12% CO2
  Other Names: S1226; CO2 Based intervention
  Arms: Standard of Care(SOC) + S-1226 at either 4% 8% or 12% CO2

SUMMARY:
This is a randomized, open-label, controlled, Phase II proof of concept study to evaluate the safety, tolerability and efficacy of S-1226 in which hospitalized subjects (n≤30) with moderate severity COVID-19 Bronchiolitis/Pneumonia will be enrolled. The safety and tolerability of S-1226 composed of PFOB with ascending doses of carbon dioxide (4%, 8%, and 12% CO2) administered twice daily will be assessed subjects in hospitalized subjects with moderate severity COVID-19 Bronchiolitis/Pneumonia.

DETAILED DESCRIPTION:
This is a randomized, open-label, controlled, Phase II proof of concept study to evaluate the safety, tolerability and efficacy of S-1226 in which hospitalized subjects with moderate severity COVID-19 Bronchiolitis/Pneumonia.

S-1226 contains a potent, safe and well-tolerated bronchodilator gas (extrinsic carbon dioxide or CO2) and perflubron (PFOB), a synthetic surfactant that facilitates restoration of surfactant function and mucus clearance. The inhaled S-1226 combination of gas, vapour and liquid aerosol penetrates obstructed airways, resulting in rapid bronchodilation, enhanced blood oxygenation, improved mucus clearance and reduction of work of breathing

The primary objective of this study is to evaluate the safety and tolerability of S-1226 composed of perflubron (PFOB) with ascending doses of carbon dioxide (4%, 8% and 12% CO2) in hospitalized subjects with moderate severity COVID-19 bronchiolitis/pneumonia. The secondary objective is to establish proof of concept that S-1226 is effective in restoring lung function in hospitalized subjects with moderate severity COVID-19 bronchiolitis/pneumonia.

The study will consist of three parts: screening period, Dosing and evaluation, follow up period.

1. During the screening period, subjects will undergo safety assessments and their eligibility to participate will be confirmed. Eligible subjects will then be randomly assigned to either the treatment arm (S-1226 + Standard of Care arm) or the non-treatment arm (Standard of Care only).
2. The dosing and evaluation period will take place over 5 days of with two doses per day. Subjects who are randomized to receive S-1226 will be started on a dose level of S-1226 (4%). If tolerated, subjects will progress from 4%, followed by 8%, and then 12%. The highest tolerated dose will then be used for the remainder of the treatment period. All doses incorporate 3mL PFOB and will be administered over a 3-4 minute treatment period. Any enrolled subject randomized to receive S-1226 will not be required to interrupt any SOC treatment which includes supplementary oxygen.

   Each S-1226 dose will be administered as inhaled gas & vapour using a Circulaire II hybrid system specifically adapted with the addition of an absolute aerosol filter installed at the site of aerosol generation. This filter removes all perflubron aerosol so that in this trial the S-1226 Gaseous Delivery System delivers an inhaled drug comprising gas (CO2 in air) and vapour (perflubron). In addition, the S-1226 Gaseous Delivery System includes a high efficiency bacterial/viral filter to scavenge any patient-generated exhaled aerosol.
3. Follow up Period will 28 days after the first dose of S1226 has been administered.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be included in the study:

  1. Male or Females between 18-80 years of age at the time of consent.
  2. Laboratory-confirmed COVID-19 infection
  3. Hospitalized for COVID-19 with clinical evidence of respiratory involvement, including at least one of the following:

     1. Symptoms/Signs: cough, respiratory distress, increased work of breathing
     2. Radiology: Chest radiograph or other chest imaging demonstrating one of bronchial thickening, increased secretions, hyperinflation, infiltrates
  4. Hypoxemia in room air, SpO2 ≤ 90%
  5. Patient belongs to one of the following two categories in the seven-point COVID-19 severity scale:

     1. Requiring supplemental oxygen by nasal prongs - Level 4 of the seven-point COVID-19 severity scale;
     2. Requiring nasal high-flow oxygen therapy,- limited to this one component of Level 5 of the seven-point COVID-19 severity scale.
  6. For women of childbearing potential involved in any sexual intercourse that could lead to pregnancy: Negative pregnancy test and willingness to use contraceptive (consistent with local regulations) during the study period.
  7. Ability to sign informed consent or, when patient is not capable of doing so, informed consent can be signed by legal/authorized representative

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Pregnant or breastfeeding females.
  2. Patients unable to receive S-1226; particularly if receiving oxygen therapy by face mask or non invasive ventilatory support
  3. Patient requires Extracorporeal Membrane Oxygenation (ECMO) and/or invasive mechanical ventilation
  4. Presence of any of the following abnormal laboratory values at screening:

     1. Absolute neutrophil count (ANC) less than 0.5 x 109 / L.
     2. Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) greater than 5 x upper limit of normal (ULN).
     3. Platelets less than 50 x109 / L.
  5. In the opinion of the investigator, progression to death is imminent and inevitable within the next 72 hours, irrespective of the provision of treatment.
  6. Subject, who in the opinion of the Investigator, is unsuitable to participate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-15 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Effects | up to 28 days
  The number and percent of treatment emergent adverse events will be monitored, recorded and graded for severity and assigned attribution. The severity will be assessed in the following manner:
  Mild: Awareness of signs or symptoms, but are easily tolerated and are of minor irritant type, causing no limitations of usual activities. Signs or symptoms may require minor action or additional therapy.
  Moderate: Discomfort severe enough to cause some limitations of usual activities and may require action or additional therapy.
  Severe: Incapacitating with inability to carry out usual activities and requires specific action and/or medical attention. Note: the term severe is not the same as "serious", which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

SECONDARY OUTCOMES:
Change in use of supplemental oxygen therapy | up to 28 days
  Measured by comparing duration in which supplemental oxygen therapy is used at baseline and after drug administration.
Normalization of body temperature, measured in degrees Celsius. | up to 28 days
  This is an exploratory efficacy measure. Assessed by a return to a normal temperature range between 36.1 and 37.2 degrees Celsius for a period of 24 hours.
Evaluation of changes in an SpO2/FiO2 ratio | up to 28 days
  This is an exploratory efficacy measure. SpO2/FiO2 ratios of 235 and 315 correlate with PaO2/FiO2 ratios of 200 for Acute Respiratory Distress Syndrome and 300 for Acute Lung Injury.
Mean change on a 7-point ordinal scale | up to 28 days
  This is an exploratory efficacy measure. The average change in points from baseline for participants in the study.
  Points 1-7 are defined below:
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalized, not requiring supplemental oxygen;
  4. hospitalized, requiring supplemental oxygen;
  5. hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both;
  6. hospitalized, requiring ECMO, invasive mechanical ventilation, or both;
  7. death.
Proportion of patients that progress to levels 6-7 of the 7-point Ordinal Scale | up to 28 days
  This is an exploratory efficacy measure. Measured by the number of participants that progress from levels 6-7.
  Points 1-7 are defined below:
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalized, not requiring supplemental oxygen;
  4. hospitalized, requiring supplemental oxygen;
  5. hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both;
  6. hospitalized, requiring ECMO, invasive mechanical ventilation, or both;
  7. death.
Time to progression to levels 6-7 of the 7-point Ordinal Scale | up to 28 days
  This is an exploratory efficacy measure. Measured by the number of days by which a change in participant ordinal score is noted.
  Points 1-7 are defined below:
  1. not hospitalized with resumption of normal activities;
  2. not hospitalized, but unable to resume normal activities;
  3. hospitalized, not requiring supplemental oxygen;
  4. hospitalized, requiring supplemental oxygen;
  5. hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both;
  6. hospitalized, requiring ECMO, invasive mechanical ventilation, or both;
  7. death.
Normalization of oxygen saturation, SpO2 > 90%, while breathing room air, sustained minimum 24 hours | up to 28 days
  This is an exploratory efficacy measure. Assessed by evaluations before and after the intervention has been administered.
Time to normalization of oxygen saturation, SpO2 > 90%, while breathing room air sustained minimum 24 hours. | up to 28 days
  This is an exploratory efficacy measure. Assessed by the duration required for oxygen saturation, SpO2, to be greater than 90%, while breathing room air and sustained for a minimum of 24 hours, following drug administration.
Change in daily symptom monitoring assessed by yes or no questions to a list of symptoms. | up to 6 days
  This is is an exploratory efficacy measure. Assessed by daily evaluations of signs and symptoms before and after the intervention has been administered.
Days of hospitalization attributable to COVID-19 disease | up to 28 days
  This is an exploratory efficacy measure. To be assessed by participants discharge date following treatment period.

OTHER OUTCOMES:
Improvement in Thoracic Imaging as assessed by a Radiologist | up to 28 days
  Following treatment evidence of change in bronchial thickening, increased secretions, hyperinflation, infiltrates will be assessed at baseline and following treatment. These include Chest X-rays and CT Scans taken during the participant's hospital stay.
Number of Participants that develop of secondary pneumonia. | up to 28 days
  To be assessed following the completion of the study.
Viral load | up to 28 days
  if available

CONTACTS AND LOCATIONS:
Overall Officials: Mark Montgomery, MD, Principal Investigator — University of Calgary
Locations (1):
- Alberta Lung Function, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swystun V, Green FHY, Dennis JH, Rampakakis E, Lalli G, Fadayomi M, Chiu A, Shrestha G, El Shahat SG, Nelson DE, El Mays TY, Pieron CA, Leigh R. A phase IIa proof-of-concept, placebo-controlled, randomized, double-blind, crossover, single-dose clinical trial of a new class of bronchodilator for acute asthma. Trials. 2018 Jun 18;19(1):321. doi: 10.1186/s13063-018-2720-6. PMID 29914544
- [Background] Green FH, Leigh R, Fadayomi M, Lalli G, Chiu A, Shrestha G, ElShahat SG, Nelson DE, El Mays TY, Pieron CA, Dennis JH. A phase I, placebo-controlled, randomized, double-blind, single ascending dose-ranging study to evaluate the safety and tolerability of a novel biophysical bronchodilator (S-1226) administered by nebulization in healthy volunteers. Trials. 2016 Jul 28;17:361. doi: 10.1186/s13063-016-1489-8. PMID 27464582
- [Background] El Mays TY, Choudhury P, Leigh R, Koumoundouros E, Van der Velden J, Shrestha G, Pieron CA, Dennis JH, Green FH, Snibson KJ. Nebulized perflubron and carbon dioxide rapidly dilate constricted airways in an ovine model of allergic asthma. Respir Res. 2014 Sep 16;15(1):98. doi: 10.1186/s12931-014-0098-x. PMID 25355286